CLINICAL TRIAL: NCT00087828
Title: Cranberry Juice Metabolites in Urine
Brief Title: Identification of the Cranberry Juice Compounds That Prevent Urinary Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: F31 AT000623-1; F31AT000623 (NIH)
Record Dates: First submitted 2004-07-14; First posted 2004-07-16 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Urinary Tract Infections
Keywords: Vaccinium macrocarpon
MeSH Terms: conditions — Urinary Tract Infections

INTERVENTIONS:
Drug: Cranberry juice cocktail

SUMMARY:
The purpose of this study is to identify the substances in cranberry juice that make it effective in reducing urinary tract infections (UTIs) in women.

DETAILED DESCRIPTION:
Urinary tract infections (UTIs) are a significant health issue, with one fourth of all women experiencing symptoms during their lifetimes. Cranberry juice has been shown to reduce the incidence of UTIs by preventing bacteria from adhering to the bladder. However, the compounds that direct this activity have not been identified. This study will identify and examine UTI-reducing compounds in cranberry juice.

Participants in this study will drink a specified amount of water following an overnight fast. Their urine will be collected 1 to 3 hours after the water is consumed. Several days later, the women will be provided with cranberry juice to replace the water in the regimen. Urine samples will be analyzed for compounds that have antibacterial or antiadhesion activity against the bacteria that cause UTIs.

ELIGIBILITY:
Inclusion Criteria:

* Good overall health

Exclusion Criteria:

* History of urinary tract infections
* Use of cranberry products or antibiotics within 1 week of study start
* Current use of any other medication
* Hypertension
* Diabetes
* Pregnancy

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5
Dates: Start 2000-11; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Susan Turner, MD, Principal Investigator — UIC
Locations (1):
- Dept Medicinal Chemistry & Pharmacognosy, COP, UIC, Chicago, Illinois, United States

REFERENCES:
- [Background] Ahuja S, Kaack B, Roberts J. Loss of fimbrial adhesion with the addition of Vaccinum macrocarpon to the growth medium of P-fimbriated Escherichia coli. J Urol. 1998 Feb;159(2):559-62. doi: 10.1016/s0022-5347(01)63983-1. PMID 9649291
- [Background] Avorn J, Monane M, Gurwitz JH, Glynn RJ, Choodnovskiy I, Lipsitz LA. Reduction of bacteriuria and pyuria after ingestion of cranberry juice. JAMA. 1994 Mar 9;271(10):751-4. doi: 10.1001/jama.1994.03510340041031. PMID 8093138
- [Background] Foo LY, Lu Y, Howell AB, Vorsa N. A-Type proanthocyanidin trimers from cranberry that inhibit adherence of uropathogenic P-fimbriated Escherichia coli. J Nat Prod. 2000 Sep;63(9):1225-8. doi: 10.1021/np000128u. PMID 11000024
- [Background] Foo LY, Lu Y, Howell AB, Vorsa N. The structure of cranberry proanthocyanidins which inhibit adherence of uropathogenic P-fimbriated Escherichia coli in vitro. Phytochemistry. 2000 May;54(2):173-81. doi: 10.1016/s0031-9422(99)00573-7. PMID 10872208
- [Background] Schmidt DR, Sobota AE. An examination of the anti-adherence activity of cranberry juice on urinary and nonurinary bacterial isolates. Microbios. 1988;55(224-225):173-81. PMID 3063927